CLINICAL TRIAL: NCT01161953
Title: Understanding the Genetic Predisposition to the Development of Primary Biliary Cirrhosis (PBC).
Brief Title: Genetic Epidemiology of Primary Biliary Cirrhosis (PBC)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Konstantinos N. Lazaridis, M.D., Hepatology Consultant, Mayo Clinic
Other Study IDs: 670-02 PBC
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Primary Biliary Cirrhosis; PBC; Cholestatic Liver Disease
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood and stool samples are collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: Genetic Analysis — Perform Genome Wide Association Studies.

SUMMARY:
Primary Biliary Cirrhosis (PBC) is a progressive liver disorder of unknown cause. Current evidence suggests that genes, the genetic material we inherit from our parents, in combination with environmental factors, likely play an important role in the development of PBC.

This study is being done to investigate whether genes make people more likely to develop PBC. Discovery of these proposed genes will help us better understand how PBC developes, and subsequently, to apply new approaches for its prevention, diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18-90 who have a history of PBC.
* PBC patients who have undergone a liver transplant are eligible.
* Family members (1st degree relatives) of enrolled PBC patients are eligible.

Exclusion Criteria:

* Individuals with no history of PBC or those unable to provide consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are patients at Mayo Clinic and are seen in the department of Gastroenterology and Hepatology are recruited by mail and carry a diagnosis of PBC. Subjects who are not Mayo Clinic patients are encouraged to contact the study coordinator by phone or email to request enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2002-03; Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Mapping of Susceptibility Genes in Adult Chronic Cholestatic Liver Diseases
  Adult chronic cholestatic liver diseases, such as Primary Biliary Cirrhosis (PBC), are progressive liver disorders of unknown cause. Current evidence suggests that genes, the genetic material we inherit from our parents, in combination with environmental factors, likely play an important role in the development of PBC.
  This study is being done to investigate whether genes (the inherited genetic material passed from parents to their children) make people more likely to develop PBC. Discovery of these proposed genes will help us to better understand how PBC progresses, and subsequently, to apply new approaches for its prevention, diagnosis and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos N Lazaridis, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lazaridis KN, Juran BD, Boe GM, Slusser JP, de Andrade M, Homburger HA, Ghosh K, Dickson ER, Lindor KD, Petersen GM. Increased prevalence of antimitochondrial antibodies in first-degree relatives of patients with primary biliary cirrhosis. Hepatology. 2007 Sep;46(3):785-92. doi: 10.1002/hep.21749. PMID 17680647
- [Background] Juran BD, Atkinson EJ, Larson JJ, Schlicht EM, Liu X, Heathcote EJ, Hirschfield GM, Siminovitch KA, Lazaridis KN. Carriage of a tumor necrosis factor polymorphism amplifies the cytotoxic T-lymphocyte antigen 4 attributed risk of primary biliary cirrhosis: evidence for a gene-gene interaction. Hepatology. 2010 Jul;52(1):223-9. doi: 10.1002/hep.23667. PMID 20578265
- [Background] Juran BD, Atkinson EJ, Larson JJ, Schlicht EM, Lazaridis KN. Common genetic variation and haplotypes of the anion exchanger SLC4A2 in primary biliary cirrhosis. Am J Gastroenterol. 2009 Jun;104(6):1406-11. doi: 10.1038/ajg.2009.103. Epub 2009 Apr 21. PMID 19491853
- [Background] Juran BD, Atkinson EJ, Schlicht EM, Fridley BL, Petersen GM, Lazaridis KN. Interacting alleles of the coinhibitory immunoreceptor genes cytotoxic T-lymphocyte antigen 4 and programmed cell-death 1 influence risk and features of primary biliary cirrhosis. Hepatology. 2008 Feb;47(2):563-70. doi: 10.1002/hep.22048. PMID 18041714
- [Background] Juran BD, Atkinson EJ, Schlicht EM, Fridley BL, Lazaridis KN. Primary biliary cirrhosis is associated with a genetic variant in the 3' flanking region of the CTLA4 gene. Gastroenterology. 2008 Oct;135(4):1200-6. doi: 10.1053/j.gastro.2008.06.077. Epub 2008 Jul 1. PMID 18778710
- [Background] Lammert C, Nguyen DL, Juran BD, Schlicht E, Larson JJ, Atkinson EJ, Lazaridis KN. Questionnaire based assessment of risk factors for primary biliary cirrhosis. Dig Liver Dis. 2013 Jul;45(7):589-94. doi: 10.1016/j.dld.2013.01.028. Epub 2013 Mar 11. PMID 23490343
- [Background] Lammert C, Juran BD, Schlicht E, Chan LL, Atkinson EJ, de Andrade M, Lazaridis KN. Biochemical response to ursodeoxycholic acid predicts survival in a North American cohort of primary biliary cirrhosis patients. J Gastroenterol. 2014 Oct;49(10):1414-20. doi: 10.1007/s00535-013-0903-1. Epub 2013 Dec 8. PMID 24317935
- [Background] Lammert C, Juran BD, Schlicht E, Xie X, Atkinson EJ, de Andrade M, Lazaridis KN. Reduced coffee consumption among individuals with primary sclerosing cholangitis but not primary biliary cirrhosis. Clin Gastroenterol Hepatol. 2014 Sep;12(9):1562-8. doi: 10.1016/j.cgh.2013.12.036. Epub 2014 Jan 16. PMID 24440215